CLINICAL TRIAL: NCT03462745
Title: Randomized Cross Over Study Comparing the First Attempt Success Rate of Intravenous Cannulation in Children Using the AccuVein AV 300 Apparatus Versus the Standard Technique
Brief Title: A Comparison of the First Attempt Success Rate of Cannulation Between the Accuvein Apparatus and Standard Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Roland Kaddoum, Associate Professor Department of Anesthesiology/ Director of Pediatric Anesthesia/ Director of Operating Room, American University of Beirut Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ANES.RK.01
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Procedural Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Cannulation with AccuVein AV 300 (Experimental): The AccuVein AV300 device helps in venepuncture and intravenous (IV) cannulation. It uses infrared light that can be absorbed by the blood hemoglobin so that veins location is clearly viewed on the skin's surface.
  Interventions: Device: AccuVein AV 300
- Standard insertion (No Intervention): Intravenous cannulation is an invasive procedure of inserting an intravenous catheter blindly through the skin, into the lumen of a peripheral vein.

INTERVENTIONS:
Device: AccuVein AV 300 — Assess the effectiveness of the AccuVein AV300 device over the standard technique in increasing the ﬁrst-time success rate (SR) for pediatric patients who needed IV cannulation
  Arms: Cannulation with AccuVein AV 300

SUMMARY:
Background: The AccuVein AV300 device helps in venepuncture and intravenous (IV) cannulation. It uses infrared light that can be absorbed by the blood hemoglobin so that veins location is clearly viewed on the skin's surface.

Objectives: To assess the effectiveness of the AV300 device over the standard technique in increasing the ﬁrst-time success rate (SR) for pediatric patients who needed IV cannulation.

Methods: This was a prospective cross study of patients aged 0-18 years scheduled for surgery or examination under anesthesia but without having an existing IV access and after providing consent form. Patients were randomized into two groups; cannulation with AV300 or standard insertion performed by experienced pediatric anesthesiologists and residents under training.

DETAILED DESCRIPTION:
Patients who fulfilled the inclusion criteria and provided informed consent were assigned to one of two groups using a randomization program that assigned research participants into group A (AccuVein AV300 assisted intravenous catheter insertion) or group B (standard technique of insertion of the intravenous cannula). After pre-anesthetic evaluation, the research participant was brought to the operating room and standard monitoring were applied (EKG, SpO2, BP) if tolerated. Anesthesia was induced via face mask with sevoflurane in 100% O2. The anesthesiologist and resident decided on a site believed to be the best for cannulation and on the size of the venous cannula as 22g or 24g. When the supervising anesthesiologist deemed it appropriate, the venous cannulation was attempted, according to the randomization groups, either with the AccuVein device (group A) or blindly (group B). A rating of the vein attempted as either difficult or easy was established by the attending anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 18 years of age, American Society of Anesthesiologist Physical Status (ASA) status I, II or III, undergoing elective surgery or examination under anesthesia, which did not have existing intravenous access.

Exclusion Criteria:

* Existing intravenous access, malformations or infections at the potential site of insertion, need for emergency surgery, and inability or unwillingness of parent or legal guardian to give written informed consent.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 184 (Actual)
Dates: Start 2013-02-10 (Actual); Primary Completion 2014-02-10 (Actual); Study Completion 2014-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland N Kaddoum, MD, Principal Investigator — American University of Beirut Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cannulation With AccuVein AV 300 | Standard Insertion
Started | 92 | 92
Completed | 92 | 92
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cannulation With AccuVein AV 300 | Standard Insertion | Total
Number analyzed (Participants) | 92 | 92 | 184
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 92 | 92 | 184
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.4 (3.2) | 4.3 (3.7) | 4.3 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 115
  Male | 35 | 34 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Lebanon | 92 | 92 | 184

OUTCOME MEASURES:

1. Primary Outcome: First Attempt Success Rates With the AccuVein 300 Device Versus Standard Method
Time Frame: Beginning of venous Cannulation until end of Cannulation, average of 1 min
Measure: Count of Participants; unit: Participants
Arm/Group | Cannulation With AccuVein AV 300 | Standard Insertion
Number analyzed (Participants) | 92 | 92
Participants | 92 | 92

ADVERSE EVENTS:
Groups:
- Cannulation With AccuVein AV 300: The AccuVein AV300 device helps in venepuncture and intravenous (IV) cannulation. It uses infrared light that can be absorbed by the blood hemoglobin so that veins location is clearly viewed on the skin's surface.
  AccuVein AV 300: Assess the effectiveness of the AccuVein AV300 device over the standard technique in increasing the ﬁrst-time success rate (SR) for pediatric patients who needed IV cannulation
  No adverse events reported.
- Standard Insertion: Intravenous cannulation is an invasive procedure of inserting an intravenous catheter blindly through the skin, into the lumen of a peripheral vein.
  No adverse events reported.
Arm/Group | Cannulation With AccuVein AV 300 | Standard Insertion
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 0/92 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes